CLINICAL TRIAL: NCT01864382
Title: Effects of the Inclusion of Exercises "Core Stability" in the Treatment of Inpatient Physiotherapy to Improve Balance in Post-stroke Patients Sitting in Subacute Phase. Randomized Clinical Trial.
Brief Title: "Core Stability" Exercises to Improve Sitting Balance in Stroke Patients
Acronym: Fisionet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rosa Cabanas Valdés (Other)
Collaborators: Corporacion Parc Tauli (Other); Institut Investigacio Sanitaria Pere Virgili (Other)
Responsible Party: Sponsor-Investigator, Rosa Cabanas Valdés, Instructor of the Physical Therapy teaching staff, Universitat Internacional de Catalunya
Organization: Universitat Internacional de Catalunya (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: UIC-FIS-2012-04
Record Dates: First submitted 2013-05-21; First posted 2013-05-29 (Estimated); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Stroke; Cerebral Stroke; Cerebrovascular Accident
Keywords: Trunk performance; exercise,; "core stability",; sitting balance
MeSH Terms: conditions — Stroke; Motor Activity | interventions — Core Stability

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Physiotherapy Exercises (Other): Standard Physiotherapy Exercises 5 days a week during 5 weeks
  Interventions: Other: Standard Physiotherapy Exercises
- Core stability (Experimental): Core stability.5 days a week during 5 weeks
  Interventions: Other: Core stability; Other: Standard Physiotherapy Exercises

INTERVENTIONS:
Other: Core stability — Core stability 5 days a week during 5 weeks
  Other Names: Trunk exercises
  Arms: Core stability
Other: Standard Physiotherapy Exercises — Standard Physiotherapy Exercises is a conventional treatment program 5 days a week during 5 weeks
  Other Names: Usual care

SUMMARY:
The stroke as cerebrovascular disease is the leading cause of permanent neurological disability and the third death in the Western world. Their affected often have motor and sensory disturbances in the form of hemiparesis with a possible influence on the balance be altered trunk muscles, important components of postural control. The treatment of stroke, covers a wide range of different strategies and approaches physiotherapy, including, specific exercises on the trunk called "core stability", performed by the patient with the help and supervision of a physiotherapist specializing in neurology, that are based on coordination, motor and proprioceptive work, especially the lumbar-pelvic. The effectiveness of these last years has been demonstrated empirically, but until now there is no sufficient evidence of the effects of these exercises on sitting balance in respect, and standing up in the subacute phase post-stroke patients. To prove the evidence raises a randomized, multicenter, blinded and where the evaluator will not participate in the analysis and processing is done by intention to treat. Patients will be divided into two groups: control (usual physiotherapy center made ) and experimental (made also 15 minutes workout "core stability"). The intervention will have a frequency of 5 days a week for 5 weeks and up to 12 weeks. The expected effect is that the experimental group patients develop better postural control at the trunk and this influences the balance in sitting, standing and walking.

DETAILED DESCRIPTION:
The deterioration in the balance sitting and poor sitting ability, clinical problems are common after stroke. These patients show a significant decrease in the performance level of the trunk, compared to healthy individuals of the same age and sex and present asymmetry of the trunk and pelvis.

Sitting involves the ability to achieve a variety of objects that are in and out of arm's length, as personal daily activities, showering, going to the bathroom and dressing. These arm movements, triggering postural adjustments in the muscles of the trunk and lower extremities, which anticipated the movement always precede the active movement. This anticipative control can be altered in subjects with stroke.

The trunk seems particularly important for balance, as stabilizes the pelvis and spine. Dean et al, (1997; 2007) and Ibrahimi (2010) showed a beneficial effect on functional scope of practice tasks, sitting in variables dynamic sitting balance, load weight of the affected side and standing. Also in the studies of Howe (2005); Verheyden (2009); Saeys (2011);Karthikbabu (2011) and Kumar (2011) with specific exercises for the trunk, favorable outcomes were obtained compared with standard treatment. However, these studies with few patients and without any monitoring, it needs to be confirmed (what is this study intended)

ELIGIBILITY:
Inclusion Criteria:

* Adults of either sex
* > 18 years with a diagnosis of stroke, ischemic or hemorrhagic origin <3 months of evolution
* Orthopedic problems not present to keep sitting. Ability to understand instructions
* The Index Barthel ˂ 70 points and Trunk Impairment Scale ˂ 16 points.

Exclusion Criteria:

* Patients with cognitive problems, Mini mental state examination ˂ 24
* Patients with a second stroke confirmed by Neurology services or previous motor disability that altered the balance, or a Rankin value not superior to 3
* The patients with stroke hemorrhagic origin with surgical treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Dynamic sitting balance | Baseline, up to 25 sessions and follow up to 24 weeks
  Trunk Impairment Scales:Is a tool to measure the motor impairment of the trunk after stroke, This scale evaluates dynamic sitting balance as well as co-ordination of trunk movement.

SECONDARY OUTCOMES:
Standing balance | Baseline, up to 25 sessions and follow up to 24 weeks
  Berg Balance Scale (BBS)assesses standing balance. This scale includes 14 common tasks of ability to maintain positions or movements of increasing difficulty by decreasing base of support from sit, to stand, to single-limb support.Each of the 14 tasks is scored on a scale from 0 (worst) to 4 (best) for a total score of 56.

OTHER OUTCOMES:
Mobility and degree of disability | Baseline, up to 25 sessions and follow up to 24 weeks
  The Barthel index is a valid scale for studying function in stroke patients.The initial Barthel score is an important prognostic factor for both recovery of function and for survival. The scale consists 10 items.

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Mª Cabanas-Valdes, Kinesiology, Principal Investigator — Universitat Internacional de Catalunya; Caritat Bagur-Calafat, Study Director — Universitat Internacional de Catalunya
Locations (2):
- Spain (2):
  - Parc Sanitari Pere Virgili, Barcelona, Catalonia
  - Consorci Hospitalari Parc Tauli, Sabadell Barcelona, Catalonia